CLINICAL TRIAL: NCT02195232
Title: Randomized, Placebo-controlled, Double-blind Phase II/III Trial of Oral Isoquercetin to Prevent Venous Thromboembolic Events in Cancer Patients.
Brief Title: Cancer Associated Thrombosis and Isoquercetin (CATIQ)
Acronym: CATIQ
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Jeffrey Zwicker, MD (Other)
Collaborators: Quercegen Pharmaceuticals (Industry); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Jeffrey Zwicker, MD, Principal Investigator, Beth Israel Deaconess Medical Center
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 14-114
Record Dates: First submitted 2014-05-13; First posted 2014-07-21 (Estimated); Results first posted 2019-11-12 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Thromboembolism of Vein VTE in Colorectal Cancer; Thromboembolism of Vein in Pancreatic Cancer; Thromboembolism of Vein in Non-small Cell Lung Cancer
Keywords: Venous Thromboembolic Events in Cancer Patients; Thromboembolism of Vein in Colorectal Cancer; Thromboembolism of Vein in Pancreatic Cancer; Thromboembolism of Vein in Non-small Cell Lung Cancer
MeSH Terms: interventions — isoquercitrin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort A - Isoquercetin (Experimental): -- Cohort A: 500 mg, Once daily, 28 days
  - For both cohorts A and B, lower extremity ultrasound will be performed at 56 days. Baseline D-dimer and correlative labs will be drawn at Day 1 and at 56 days. Patients will be followed for survival after completion of 56 days.
  Interventions: Drug: Isoquercetin
- Cohort B - Isoquercetin (Experimental): --Cohort B: 1000 mg, Once daily, 28 days
  - For both cohorts A and B, lower extremity ultrasound will be performed at 56 days. Baseline D-dimer and correlative labs will be drawn at Day 1 and at 56 days. Patients will be followed for survival after completion of 56 days.
  Interventions: Drug: Isoquercetin

INTERVENTIONS:
Drug: Isoquercetin
  Other Names: quercetin-3-O-glucoside; 482-35-9

SUMMARY:
This research study is evaluating a drug called isoquercetin to prevent venous thrombosis (blood clots), in participants who have pancreas, non small cell lung cancer or colorectal cancer.

DETAILED DESCRIPTION:
* This research study is a Phase II/III clinical trial.

  --The goal of this trial is to evaluate if isoquercetin can prevent blood clots in patients with pancreas, non small cell lung cancer or colorectal cancer. In the Phase II part of this study, the investigators are looking for the dose of isoquercetin to reduce D-dimer and demonstrate safety.
* Phase III Endpoint and Treatment Plan

  * Primary Endpoint for Phase III portion of protocol: Cumulative incidence of VTE.
  * Following the completion of the phase II portion, enrolled patients will be randomized 1:1 to Arm C (isoquercetin) or Arm D (placebo). The dose for Arm C will be determined after evaluation of the Phase II portion of the trial. The protocol will be amended when the decision is made whether to proceed to Phase III and what dose to use for Arm C. The study will be double-blinded to treatment arm. Lower extremity ultrasound will be performed at 56 days. Baseline D-dimer and correlative labs will be drawn at Day 1 and at 56 days. Patients will be followed for survival after completion of 56 days.
  * At BIDMC, optional blood draw will be performed at time 0 and 4 hours following the first dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet the following criteria on screening examination to be eligible to participate in phase 2 and 3 of the study:
* Participants must have histologically confirmed malignancy that is metastatic or currently unresectable.
* Eligible malignancies include:

  * Adenocarcinoma of the pancreas (currently unresectable or metastatic)
  * Colorectal (stage IV)
  * Non-small cell lung cancer (currently unresectable stage III or stage IV)
* Receiving or scheduled to receive first or second line chemotherapy (within 30 days of registration)
* Minimum age 18 years. Because limited dosing or adverse event data are currently available on the use of isoquercetin in participants <18 years of age, children are excluded from this study but will be eligible for future pediatric isoquercetin trials.
* Life expectancy of greater than 4 months.
* ECOG performance status ≤2 (see Appendix B ).
* Patient must be able to swallow capsules (phase III only)
* Participants must have preserved organ and marrow function as defined below:

  * Absolute neutrophil count ≥1,000/mcL
  * Platelets ≥ 90,000/mcL
  * PT and PTT ≤ 1.5 x upper limit of normal
  * Total bilirubin < 2.0 mg/dl
  * AST (SGOT)/ALT (SGPT) ≤ 2.5 X institutional upper limit of normal Creatinine < 2.0 mg/dl
* The effects of isoquercetin on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants may not be receiving any other study agents.
* Participants with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Prior history of documented venous thromboembolic event within the last 2 years (excluding central line associated events whereby patients completed anticoagulation).
* Active bleeding or high risk for bleeding (e.g. known acute gastrointestinal ulcer)
* History of significant hemorrhage (requiring hospitalization or transfusion) outside of a surgical setting within the last 24 months
* Familial bleeding diathesis
* Known diagnosis of disseminated intravascular coagulation (DIC)
* Currently receiving anticoagulant therapy
* Current daily use of aspirin (>81mg daily), Clopidogrel (Plavix), cilostazol (Pletal), aspirin-dipyridamole (Aggrenox) (within 10 days) or considered to use regular use of higher doses of non-steroidal anti-inflammatory agents as determined by the treating physician (e.g ibuprofen > 800 mg daily or equivalent).
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Known intolerance of niacin or ascorbic acid (including known G6PD deficiency)
* Pregnant women are excluded from this study because isoquercetin is a PDI inhibitor with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk of adverse events in nursing infants secondary to treatment of the mother with isoquercetin, breastfeeding should be discontinued if the mother is treated with isoquercetin. These potential risks may also apply to other agents used in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Zwicker, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (11):
- United States (11):
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - VA Northern California Health Care System, Sacramento, California
  - VA Connecticut Healthcare System, West Haven, Connecticut
  - Veterans Affair Medical Center, Washington D.C., District of Columbia
  - York Hospital-Oncology Treatment Center, York Village, Maine
  - Boston VA Healthcare System, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mount Auburn Hospital, Waltham, Massachusetts
  - Washington University in St. Louis, St Louis, Missouri
  - Providence VA Medical Center, Providence, Rhode Island
  - White River Junction VA Medical Center, White River Junction, Vermont

REFERENCES:
- [Derived] Zwicker JI, Schlechter BL, Stopa JD, Liebman HA, Aggarwal A, Puligandla M, Caughey T, Bauer KA, Kuemmerle N, Wong E, Wun T, McLaughlin M, Hidalgo M, Neuberg D, Furie B, Flaumenhaft R; CATIQ Investigators11. Targeting protein disulfide isomerase with the flavonoid isoquercetin to improve hypercoagulability in advanced cancer. JCI Insight. 2019 Feb 21;4(4):e125851. doi: 10.1172/jci.insight.125851. eCollection 2019 Feb 21. PMID 30652973

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A (Isoquercetin 500 mg): Patients will receive isoquercetin 500 mg once daily (2 capsules).
- Cohort B (Isoquercetin 1000 mg): Patients will receive isoquercetin 1000 mg once daily (4 capsules).
Period: Overall Study
Arm/Group | Cohort A (Isoquercetin 500 mg) | Cohort B (Isoquercetin 1000 mg)
Started | 32 (patients consented) | 32 (patients consented)
Completed | 28 (Evaluated for VTE and safety) | 29 (Evaluated for VTE and safety)
Not Completed | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A (Isoquercetin 500 mg) | Cohort B (Isoquercetin 1000 mg) | Total
Number analyzed (Participants) | 32 | 32 | 64
Age, Categorical [Count of Participants; unit: Participants] — Population: Evaluated for VTE and safety
  Participants
    number analyzed (Participants) | 28 | 29 | 57
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 15 | 17 | 32
    >=65 years | 13 | 12 | 25
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Evaluated for VTE and safety
  Participants
    number analyzed (Participants) | 28 | 29 | 57
    Female | 14 | 9 | 23
    Male | 14 | 20 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Evaluated for VTE and safety
  Participants
    number analyzed (Participants) | 28 | 29 | 57
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 2 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 4 | 5 | 9
    White | 23 | 19 | 42
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Count of Participants; unit: Participants] — Population: Evaluated for VTE and safety
  Participants
    United States: number analyzed (Participants) | 28 | 29 | 57
    United States | 28 | 29 | 57

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in D-dimer Value
Description: D-dimer concentrations will be compared for each patient at day 0 and day 56 by a paired-t test analysis. Analysis will be performed on an intention to treat basis for patients who undergo randomization and completed the baseline and day 56 D-dimer assessments.
Time Frame: Baseline, 56 Day
Population: The analysis data set is comprised of evaluable patients.
Measure: Median (Full Range); unit: percent change
Arm/Group | Cohort A (Isoquercetin 500 mg) | Cohort B (Isoquercetin 1000 mg)
Number analyzed (Participants) | 28 | 29
percent change | 9.9 [-51.1 to 74.2] | -21.9 [-63.3 to 36.5]
Statistical Analysis 1: Comparison: Cohort A (Isoquercetin 500 mg) vs Cohort B (Isoquercetin 1000 mg); Test type: Other; p = 0.92, t-test, 2 sided

2. Secondary Outcome: Number of Participants With Hemorrhage
Description: Investigating the safety of isoquercetin in cancer patients
Time Frame: study visits until day 56
Measure: Count of Participants; unit: Participants
Groups:
- Cohort A (Isoquercetin 500 mg): Cohort A: Patients will receive isoquercetin 500 mg once daily (2 capsules) for 28 days.
  Lower extremity ultrasound will be performed at 56 days. Baseline D-dimer and correlative labs will be drawn at Day 1 and at 56 days. Patients will be followed for survival after completion of 56 days.
- Cohort B (Isoquercetin 1000 mg): Cohort B: Patients will receive isoquercetin 1000 mg once daily (4 capsules) for 28 days.
  Lower extremity ultrasound will be performed at 56 days. Baseline D-dimer and correlative labs will be drawn at Day 1 and at 56 days. Patients will be followed for survival after completion of 56 days.
Arm/Group | Cohort A (Isoquercetin 500 mg) | Cohort B (Isoquercetin 1000 mg)
Number analyzed (Participants) | 28 | 29
Participants | 2 | 2

3. Secondary Outcome: Cumulative Incidence of VTE at 56 Days
Description: To investigate the cumulative incidence of VTE according to tissue factor bearing microparticle status (and isoquercetin randomization).
Time Frame: 56 days
Population: All patients who began assigned treatment were analyzed.
Measure: Number; unit: participants
Groups:
- Cohort A - Isoquercetin: -- Cohort A: 500 mg, Once daily, 28 days
  - For both cohorts A and B, lower extremity ultrasound will be performed at 56 days. Baseline D-dimer and correlative labs will be drawn at Day 1 and at 56 days. Patients will be followed for survival after completion of 56 days.
  Isoquercetin
- Cohort B - Isoquercetin: --Cohort B: 1000 mg, Once daily, 28 days
  - For both cohorts A and B, lower extremity ultrasound will be performed at 56 days. Baseline D-dimer and correlative labs will be drawn at Day 1 and at 56 days. Patients will be followed for survival after completion of 56 days.
  Isoquercetin
Arm/Group | Cohort A - Isoquercetin | Cohort B - Isoquercetin
Number analyzed (Participants) | 28 | 29
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: All adverse events data were collected form the time of the first dose (Day 1) of study treatment, through the study and until the final study visit (Day 56).
Description: All serious adverse events that occur after the initial dose of study treatment, during treatment, or within 30 days of the last dose of treatment must be reported to the Overall Principal Investigator.
Arm/Group | Cohort A (Isoquercetin 500 mg) | Cohort B (Isoquercetin 1000 mg)
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/29
Other Adverse Events (participants affected / at risk) | 11/28 | 3/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (Isoquercetin 500 mg) (N=28) | Cohort B (Isoquercetin 1000 mg) (N=29)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Gastroesophageal reflux (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Weight loss (Investigations) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrointestinal (Gastrointestinal disorders) | 0 (0) | 2 (2) — Lower gastrointestinal hemorrhage

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-27): https://cdn.clinicaltrials.gov/large-docs/32/NCT02195232/Prot_SAP_000.pdf